CLINICAL TRIAL: NCT01865708
Title: Pilot Study of the Safety of a Daily Ethanol Lock for Urinary Catheters in Critically Ill Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Jana Stockwell, M.D., Children's Healthcare of Atlanta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ethanol Lock, Safety
Record Dates: First submitted 2013-05-09; First posted 2013-05-31 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Complication of Urinary Catheter
Keywords: Ethanol Lock; Alcohol lock; Urinary catheter; Safety
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ethanol lock (Other): Ethanol lock, utilizing 74% ethanol, will begin within 24 hours of urinary catheter placement. The lock will be done every 24 hours for 1 hour. The volume that will be instilled depends upon the fill volume of the catheter, which is imprinted by the manufacturer on each catheter. Once the alcohol is in the catheter, the proximal end of the catheter will be clamped for 1 hour. After the 1 hour dwell time, the clamp will be removed and the alcohol in the lumen of the catheter will be flushed out by the patient's own urine output.
  Interventions: Drug: Ethanol Lock

INTERVENTIONS:
Drug: Ethanol Lock — Ethanol lock, utilizing 74% ethanol, will begin within 24 hours of urinary catheter placement. The lock will be done every 24 hours for 1 hour. The volume that will be instilled depends upon the fill volume of the catheter, which is imprinted by the manufacturer on each catheter. Once the alcohol is in the catheter, the proximal end of the catheter will be clamped for 1 hour. After the 1 hour dwell time, the clamp will be removed and the alcohol in the lumen of the catheter will be flushed out by the patient's own urine output.
  Other Names: Ethanol; Dehydrated alcohol

SUMMARY:
Hypothesis 1: Blood alcohol concentration will be <25 mg/100ml (equivalent to a blood alcohol concentration of <0.025%) after a 1 hour urinary catheter ethanol lock.

Hypothesis 2: Daily urinary catheter ethanol locks will not result in increased hematuria or increased urinary white cells.

DETAILED DESCRIPTION:
This study involves a confirmatory/refuting approach to the above stated hypothesis. The investigators will test this hypothesis by addressing the following aims/objectives:

Specific Aim 1:

Quantify blood alcohol levels after a 1 hour 74% ethanol lock in urinary catheters utilized in the Pediatric Intensive Care Unit.

Specific Aim 2:

Compare cellular components in urinalyses after the introduction of the ethanol locks.

Potential study subjects will be recruited from the Children's Healthcare of Atlanta - Egleston Pediatric Intensive Care Unit. Children that are anticipated to have an indwelling urinary catheter for >48 hours will be included. For this pilot study, the investigators will enroll 10 patients. Subject ages will range from 6 months to 17 years. Children who are on a service other than Critical Care Medicine will have clearance from the primary team prior to approaching for enrollment. The consent process will take place prior to or during the initial 24 hours of urinary catheter placement.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months - 17 years
* Urinary catheter placed at Children's Healthcare of Atlanta
* Anticipated urinary catheter need for > 48 hours
* Parent or legal guardian (or patient when applicable) consent for enrollment.

Exclusion Criteria:

* 18 yo or older.
* Urosepsis at time of study enrollment
* Known bladder or genitourinary abnormalities
* Chronic bladder drainage regimen
* Urologic surgeries (as part of the current admission)
* Medical urgency preventing timely administration of the consenting process, or any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating.
* Anuria or oliguria (<0.5 cc/kg/hr averaged over the previous 12 hours)
* Other technical considerations that would prevent the timely acquisition of sufficient samples such as (but not limited to) absence of a study team member.
* Parent or legal guardian (or patient when applicable) refuses to sign informed consent.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jana A Stockwell, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Helathcare of Atlanta at Egleston, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teppa BE, Stockwell JA. Safety of daily ethanol locks for urinary catheters in critically ill children: a pilot study. Am J Infect Control. 2015 Oct 1;43(10):1114-5. doi: 10.1016/j.ajic.2015.05.012. Epub 2015 Jun 19. PMID 26099520

RESULTS

PARTICIPANT FLOW:
Groups:
- Ethanol Lock: 74% Ethanol lock will begin within 24 hours of urinary catheter placement. Lock will be done every 24 hours for 1 hour. The volume that will be instilled depends upon the fill volume of the catheter, which is imprinted by the manufacturer on each catheter. Once the alcohol is in the catheter, the proximal end of the catheter will be clamped for 1 hour. After 1 hour dwell time, the clamp will be removed and catheter will be flushed out by the patient's own urine output.
Period: Overall Study
Arm/Group | Ethanol Lock
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ethanol Lock
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.7 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Blood Alcohol Level
Description: An ethanol lock, utilizing 74% ethanol, will begin within 24 hours of catheter placement. The lock will be done every 24 hours for 1 hour. Blood alcohol levels will be obtained every day, approximately 1 hour after ethanol lock release, for 3 days: at baseline, 1 day post catheter placement, 2 days post catheter placement, and 3 days post catheter placement. Number of participants with Blood Alcohol Levels exceeding 10 mg/100 ml on any study day was analyzed.
Time Frame: up to 3 days
Population: Number of patients with detectable blood alcohol level, defined as >= 10 mg/dL.
Measure: Count of Participants; unit: Participants
Arm/Group | Ethanol Lock
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Urine Analysis
Description: An ethanol lock, utilizing 74% ethanol, will begin within 24 hours of catheter placement. The lock will be done every 24 hours for 1 hour, for a total of 3 days.
  A baseline urinalysis will be obtained prior to the first instillation of ethanol, looking for hematuria.
  A urinalysis will be obtained approximately 1 hour after the lock is released. Data shown is the mean increase in red blood cells per high powered field after ethanol instillation averaged across all post-ethanol lock days and all patients compared to the mean baseline red blood cells per high powered field in urinalysis prior to any ethanol lock.
Time Frame: Data shown is the mean increase in red blood cells per high powered field after ethanol instillation averaged across all post-EL days and all patients compared to the mean baseline red blood cells per high powered field in urinalysis prior to any EL.
Population: Change in detectable red blood cells per high powered field in urinalysis. Data shown is the mean increase in red blood cells per high powered field after ethanol instillation averaged across all post-EL days and all patients compared to the mean baseline red blood cells per high powered field in urinalysis prior to any EL.
Measure: Mean (Standard Deviation); unit: red blood cells per high powered field
Arm/Group | Ethanol Lock
Number analyzed (Participants) | 10
red blood cells per high powered field | 90.1 (226.4)

ADVERSE EVENTS:
Arm/Group | Ethanol Lock
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethanol Lock (N=10)
Microscopic hematuria (Renal and urinary disorders) | 4 (5) — Microscopic hematuria (>100 RBC/HPF) detected by lab analysis of urine specimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No